CLINICAL TRIAL: NCT07389733
Title: Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HRS-6208 in Combination With HRS-8080 ± HRS-6209, or in Combination With Fulvestrant ± HRS-6209, or in Combination With Letrozole ± HRS-6209 in Patients With Advanced Unresectable or Metastatic Breast Cancer: an Open Label, Multicenter, Phase Ib/II Study
Brief Title: A Study of HRS-6208 in Combination With HRS-8080, or Fulvestrant, or Letrozole, With or Without HRS-6209 in Patients With Advanced Unresectable or Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-6208-201-BC
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Advanced Unresectable or Metastatic Breast Cancer of Adults
MeSH Terms: interventions — Fulvestrant; Letrozole

STUDY DESIGN:
Intervention Model Description: An open label, multicenter, phase Ib/II study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: HRS-6208 + HRS-8080 ± HRS-6209 (Experimental): HRS-6208 + HRS-8080 ± HRS-6209.
  Interventions: Drug: HRS-6208 Capsule; Drug: HRS-6209 Capsule; Drug: HRS-8080 Tablet
- Arm B: HRS-6208 + Fulvestrant ± HRS-6209 (Experimental): HRS-6208 + Fulvestrant ± HRS-6209.
  Interventions: Drug: HRS-6208 Capsule; Drug: HRS-6209 Capsule; Drug: Fulvestrant injection
- Arm C: HRS-6208 + Letrozole ± HRS-6209 (Experimental): HRS-6208 + Letrozole ± HRS-6209.
  Interventions: Drug: HRS-6208 Capsule; Drug: HRS-6209 Capsule; Drug: Letrozole tablets

INTERVENTIONS:
Drug: HRS-6208 Capsule — HRS-6208 capsule.
Drug: HRS-6209 Capsule — HRS-6209 capsule.
Drug: HRS-8080 Tablet — HRS-8080 tablet.
  Arms: Arm A: HRS-6208 + HRS-8080 ± HRS-6209
Drug: Fulvestrant injection — Fulvestrant injection.
  Arms: Arm B: HRS-6208 + Fulvestrant ± HRS-6209
Drug: Letrozole tablets — Letrozole tablets.
  Arms: Arm C: HRS-6208 + Letrozole ± HRS-6209

SUMMARY:
This study aims to evaluate the safety, tolerability, efficacy and pharmacokinetics of HRS-6208 in combination with HRS-8080 ± HRS-6209, or in combination with fulvestrant ± HRS-6209, or in combination with letrozole ± HRS-6209 in patients with advanced unresectable or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 18-75 (inclusive);
2. ECOG score 0-1;
3. Estimated survival time ≥ 12 weeks;
4. Possessing adequate bone marrow and organ function;
5. Participants of reproductive/childbearing potential must agree to take adequate and effective contraceptive measures from the time they sign the informed consent form, during the study treatment period, and up to 2 years after the last use of the trial medication;
6. Participants must provide informed consent for this study before the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Within 5 years prior to the first dose of study medication, the occurrence of other malignancies, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, and post-radical surgery thyroid papillary carcinoma;
2. Active brain metastasis, carcinomatous meningitis, spinal cord compression, or history of primary central nervous system tumors;
3. Severe bone damage caused by tumor bone metastasis as determined by the investigator;
4. Adverse events caused by previous anti-tumor treatment have not been resolved;
5. Participants with one of multiple factors affecting oral medication;
6. History of severe cardiovascular and cerebrovascular diseases;
7. Presence of severe infections;
8. Significant clinically meaningful bleeding within 3 months prior to the first dose of study medication;
9. Active autoimmune diseases, history of immune deficiency, history of autoimmune diseases, or history of diseases or syndromes requiring systemic steroid hormone or immunosuppressive drug treatment, or acquired conditions (HIV infection), congenital immune deficiency diseases, or history of organ transplantation;
10. Active untreated hepatitis;
11. History of active tuberculosis infection within 1 year prior to enrollment, or history of active tuberculosis infection more than 1 year ago without standard treatment;
12. Washout period of prior drug or treatment did not meet protocol requirements before the first dose of study medication;
13. Prior use of prohibited drugs specified in the protocol;
14. Is pregnant or breastfeeding or planning to become pregnant within 2 years after the last dose of study medication;
15. History of clear neurological or psychiatric disorders, and participants with a history of psychiatric drug abuse or drug addiction;
16. Allergic reactions to any study drug or excipients;
17. Factors confirmed by the investigator as unsuitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | The DLT will be evaluated for the last participant in each dose group 28 days after the first dose.
Recommended phase II dose (RP2D) | The evaluation of RP2D will be completed approximately one year later than DLT evaluation.
Incidence and severity of adverse events (AEs) | Each individual participant will be followed for approximately 8 months, and the entire study process will last for approximately 36 months.
Objective response rate (ORR) | For a single subject, the duration will be approximately 8 months, while the entire research process will last for 36 months.

SECONDARY OUTCOMES:
Disease control rate (DCR) | The duration for a single subject will be approximately 8 months, and the entire research process will last for 36 months.
Duration of response (DoR) | The duration for a single subject will be approximately 8 months, and the entire research process will last for 36 months.
Progression-free survival (PFS) | The duration for a single subject will be approximately 8 months, and the entire research process will last for 36 months.
Overall survival (OS) | The duration for a single subject will be approximately 8 months, and the entire research process will last for 36 months.
The blood drug concentration of HRS-6208 | The duration for a single subject will be approximately 8 months, and the entire research process will last for 36 months.
The blood drug concentration of HRS-8080 | The duration for a single subject will be approximately 8 months, and the entire research process will last for 36 months.
The blood drug concentration of HRS-6209 | The duration for a single subject will be approximately 8 months, and the entire research process will last for 36 months.
The blood drug concentration of Letrozole | The duration for a single subject will be approximately 8 months, and the entire research process will last for 36 months.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided